CLINICAL TRIAL: NCT03839069
Title: The Effects of Minor Salivary Gland Transplantation for Cicatrizing Conjunctivitis
Brief Title: Minor Salivary Gland Transplantation for Cicatrizing Conjunctivitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201503027DINB
Record Dates: First submitted 2016-08-31; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Cicatrizing Conjunctivitis; Stevens-Johnson Syndrome Toxic Epidermal Necrolysis Spectrum; Sjogren Syndrome; Mucous Membrane Pemphigoid; Chronic Graft Versus Host Disease; Chemical Burn to Eye
MeSH Terms: conditions — Stevens-Johnson Syndrome; Sjogren's Syndrome; Pemphigoid, Benign Mucous Membrane; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minor Salivary Gland Transplantation (Experimental): Cicatrizing conjunctivitis patients that received minor salivary gland transplantation for dry eye treatment.
  Interventions: Procedure: minor salivary gland transplantation

INTERVENTIONS:
Procedure: minor salivary gland transplantation — The investigators will harvest the autologous labial salivary gland tissue and transplant to the upper and lower conjunctival fornix of the lesion eye.

SUMMARY:
This is a prospective study that aimed to observe the therapeutic effects of minor salivary gland transplantation for cicatrizing conjunctivitis patients.

DETAILED DESCRIPTION:
Cicatrizing conjunctivitis can be the common presentation of many ocular surface diseases as Stevens-Johnson syndrome (SJS), mucous membrane pemphigoid (MMP), chemical burn, Sjogren syndrome, chronic graft-versus-host disease (GVHD) and ocular trauma. Ocular dryness in combination with symblepharon and corneal opacity in these patients could lead to the poor visual and life quality, and less favorable prognosis of ocular reconstruction.

This study aims to prospectively evaluate the therapeutic effects of minor salivary gland transplantation for cicatrizing conjunctivitis. The investigators evaluate the saliva-tear productivity (functional outcome) and the survival of graft (anatomical outcome) every three months. The investigators would also validate whether minor salivary gland transplantation is beneficial for the participant prior to further ocular reconstruction as limbal transplantation and corneal grafting.

ELIGIBILITY:
Inclusion Criteria:

* age 20-85 years old
* unilateral or bilateral cicatrizing conjunctivitis
* severe aqueous deficiency dry eye ( Schirmer I test result of less than 2mm)
* chronic ocular surface disease score (COCS) over 3 points
* Oxford scheme over grade III

Exclusion Criteria:

* active ocular infection
* active corneal melting
* severe xerostomia (modified Schirmer I test result of less than 25mm)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
the change of Schirmer's test result (basic tear secretion in mm) from baseline to 12 months after operation | the Schirmer's test will be performed every three months until 12 months after operation
  to compare the Schirmer's test between baseline and 12 months after operation. The higher Schirmer's test results, the better tear secretion function.
the change of ocular surface disease index (OSDI) ( ranged from 0-100) from baseline to 12 months after operation | the OSDI will be monitored every three months until 12 months
  to compare the OSDI between baseline and 12 months after operation. The higher the OSDI value, the worse of subjective ocular surface disease related symptoms.
the change of chronic ocular complication score (COCS) ( ranged from 0-12) from baseline to 12 months after operation | the COCS will be monitored every three months until 12 months after operation
  to compare the COCS between baseline and 12 months after operation. The higher the COCS scores, the more ocular surface complications.

SECONDARY OUTCOMES:
the change of conjunctival impression cytology scores (ranged from 0-5) from baseline to 12 months after operation | the impression cytology will be performed every three months until 12 months after operation
  to compare the scores of conjunctival impression cytology between baseline and 12 months after operation. The higher the conjunctival impression cytology scores, the worse squamous metaplasia of the ocular surface.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Sang Chu, MD, MS, Principal Investigator — Department of Ophthalmology, NTUH
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
for research purpose only